CLINICAL TRIAL: NCT03074981
Title: Novel Methods for Management of Complicated Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-3907-17-SMC
Record Dates: First submitted 2017-02-23; First posted 2017-03-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Complications Wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined TopClosure & Vcare Alpha Treatment (Experimental): The investigators will debride the wound if necessary. Wound biopsies will be taken to determine the existing pathogens and direct the antibiotic treatment.
  Wound measurements will be taken. Afterwards the wound will be approximated by the TopClosure device and the patient will be connected to a Negative Wound pressure device Vcare Alpha.
  The investigators will change dressings according to schedule. If the wound is clean the investigators will change dressings every 3-5 days, If the wound is infected the investigators will change dressings every 2-4 days, If the investigators encounter a severe infected wound with a lot of pus the investigators will change dressings every 1-3 days, The investigators will determine the time to heal when the wound is clean and there is no further need for Negative Pressure Wound Treatment (ROI-NPT) up to 10 weeks.
  Interventions: Device: Combined TopClosure & Vcare Alpha

INTERVENTIONS:
Device: Combined TopClosure & Vcare Alpha — Combined TopClosure & Vcare Alpha Treatment. The investigators will debride the wound if necessary. Wound biopsies will be taken to determine the existing pathogens and direct the antibiotic treatment.
  Wound measurements will be taken. Afterwards the wound will be approximated by the TopClosure device and the patient will be connected to a Negative Wound pressure device Vcare Alpha.
  The investigators will change dressings according to schedule. If the wound is clean the investigators will change dressings every 3-5 days, If the wound is infected the investigators will change dressings every 2-4 days, If the investigators encounter a severe infected wound with a lot of pus the investigators will change dressings every 1-3 days, The investigators will determine the time to heal when the wound is clean and there is no further need for Negative Pressure Wound Treatment (ROI-NPT) up to 10 weeks.

SUMMARY:
Difficult to heal wounds are a common and complex medical problem, causing suffer to the patients and challenging medical, social and economic burden on the health system. Based on data from the western world, it is estimated that in Israel, at any given time, 30 to 60 thousand patients with difficult to heal wounds. Among diabetics patients, it is estimated that 15% to 25% will develop a difficult to heal foot wounds during their live time.

The medical definition of a difficult to heal wounds is: a wound showing no signs of recovery after 4-6 weeks of treatment. Most of these wounds are caused by anaerobic bacteria inventions.

One of the methods for the treatment of difficult to heal wounds is - ROI-RNPT (Regulated Oxygen -Enriched & Irrigation Negative Pressure -Assisted Wound Therapy).

This method creates in the wound a negative pressure in the presence of oxygen and irrigation applied directly into the wound bed.

As part of the wound closure process the investigators will use the "external tissue expansion". This method under clinical use is exercised by the - "Top Closure" "tension relief system" (TRS).

In this study, the investigators intend to investigate whether ROI-NPT system combined with TopClosure, is effective for the treatment of difficult to heal wounds, compared with methods currently in use.

DETAILED DESCRIPTION:
1. The investigators will debride the wound if necessary. Wound biopsies will be taken to determine the existing pathogens and direct the antibiotic treatment.
2. Wound measurements will be taken (Width, length and depth).
3. Afterwards the wound will be closed with the TopClosure device and the patient will be connected to a Negative Wound pressure device Vcare Alpha.
4. the investigators will change dressings according to schedule. If the wound is clean the investigators will change dressings every 3-5 days. If the wound is infected the investigators will change dressings every 2-4 days. If the investigators encounter a severe infected wound with a lot of pus the investigators will change dressings every 1-3 days.
5. the investigators will determine the time to heal when the wound is clean and there is no further need for Negative Pressure Wound Treatment (ROI-NPR) up to 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1.A patient in our in-patient rehabilitation ward that is willing to participate in our study and is willing to be constrained to his bed for the time of the study.

Exclusion Criteria:

1. Patient with cognitive impairments interfering with his or her ability to understand the instructions by our team.
2. Patient that is not willing to be constrained to his bed for the time of the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Time to wound healing | determine the time to heal from connecting the patient to the Vcare Alpha device until the wound is clean and there is no further need for Negative Pressure Wound Treatment up to 10 weeks
  the wound will be closed with the TopClosure device and the patient will be connected to a Negative Wound pressure device Vcare Alpha.

CONTACTS AND LOCATIONS:
Overall Officials: Sheba Medical Center, Principal Investigator — medical center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Topaz, M., Bisker, O., Litmanovitch, M., & Keren, G. Application of regulated oxygen-enriched negative pressure-assisted wound therapy in combating anaerobic infections. European Journal of Plastic Surgery, 34(5), 351-358, 2011
- [Result] Topaz M, Carmel NN, Topaz G, Zilinsky I. A substitute for skin grafts, flaps, or internal tissue expanders in scalp defects following tumor ablative surgery. J Drugs Dermatol. 2014 Jan;13(1):48-55. PMID 24385119